CLINICAL TRIAL: NCT07200024
Title: Virtual Functional- Based Treadmill Training on Gait Parameters in Subacute Stroke Patients: A Randomized Control Trial
Brief Title: Virtual Functional- Based Treadmill Training on Gait Parameters in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: gait training
Record Dates: First submitted 2025-09-10; First posted 2025-09-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Gait Biomechanics
Keywords: Virtual functional- based treadmill; gait parameters; subacute stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Virtual functional- based treadmill training
  Interventions: Other: Virtual functional- based treadmill training
- control group (Active Comparator): gait training for stroke patients
  Interventions: Other: gait training

INTERVENTIONS:
Other: Virtual functional- based treadmill training — rehabilitation technique that combines virtual reality (VR) with treadmill training to improve gait, balance, and functional mobility for individuals with conditions like stroke
  Arms: study group
Other: gait training — a specialized form of physical therapy focused on improving a person's walking ability, balance, and coordination after an injury, stroke, neurological condition, or other illness.
  Arms: control group

SUMMARY:
A significant of this study to determine effect of Virtual functional- based treadmill training on gait parameters in patients after stroke

ELIGIBILITY:
Inclusion Criteria:

* duration of illness 6 months
* grade 1+ modified ashower scale
* circumduction gait

Exclusion Criteria:

* spasticity more than grade 2
* dependent patients

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
gait prameters | 4 weeks
  Basic spatiotemporal parameters
  1. step time,
  2. stride time,
  3. swing time
  4. stride length
  5. velocity
  6. srtide lenght were extracted from all systems by 2D camera

CONTACTS AND LOCATIONS:
Locations (1):
- Al Zaytoonah University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No